CLINICAL TRIAL: NCT01413412
Title: Full-thickness Skin vs. Synthetic Mesh in the Repair of Large Incisional Hernia - a Prospective Randomized Controlled Study
Brief Title: Full-thickness Skin vs. Synthetic Mesh in the Repair of Large Incisional Hernia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Leonard Clay, Doctor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2009/227-31/3
Record Dates: First submitted 2011-08-09; First posted 2011-08-10 (Estimated); Last update posted 2015-09-29 (Estimated); Status verified 2015-09

CONDITIONS: Ventral Hernia; Postoperative Pain
Keywords: Ventral Hernia; Postoperative Pain; Ventral Hernia Pain Questionnaire; Postoperative Abdominal wall and muscle function; Biodex
MeSH Terms: conditions — Hernia, Ventral; Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hernia repair using full-thickness skin graft (Experimental): 25 patients
  Interventions: Procedure: Ventral hernia repair using full thickness skin graft
- Hernia repair using Mesh (Experimental): 25 patients
  Interventions: Procedure: Ventral hernia repair using mesh

INTERVENTIONS:
Procedure: Ventral hernia repair using full thickness skin graft — 25 patients
  Arms: Hernia repair using full-thickness skin graft
Procedure: Ventral hernia repair using mesh — 25 patients
  Arms: Hernia repair using Mesh

SUMMARY:
This is a prospective randomized study to compare surgical methods for the repair of large abdominal hernia.

DETAILED DESCRIPTION:
Patients with giant (>10 cm in diameter) abdominal wall hernia are included in a prospective randomized study comparing conventional mesh repair with the best possible method to onlay full thickness skin grafts.

ELIGIBILITY:
Inclusion Criteria:

* ventral hernia > 10 centimeters, abdominal wall pain or discomfort, desire hernia repair.

Exclusion Criteria:

* < 18 years of age, ongoing pregnancy or nursing, ongoing immunosuppressive treatment,ongoing smoking.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2009-12; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Rate of complication | 3 month, 1 year and 3 year post-operative clinical follow-up
  Complications will be assessed over a 3 year period of regular follow-up by an objective surgeon who is unaware of which surgical method which was used. Eventual complications may include infection, bleeding, seroma and fistula formation.

SECONDARY OUTCOMES:
Ventral Hernia Pain Questionnaire (VHPQ) | 1 year period of follow-up
  All subjects will complete the VHPQ which will be used to assess their pre- and postoperative pain.
Abdominal wall function | 3 year period of follow up
  All subjects will undergo testing of abdominal wall function and strength using the Biodex.

CONTACTS AND LOCATIONS:
Overall Officials: Karin Strigård, MD, Study Director — Karolinska Institute CLINTEC; Leonard Clay, MD, Principal Investigator — Karolinska Institute CLINTEC; Ulf Gunnarsson, MD, Study Chair — Karolinska Institute CLINTEC
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden

REFERENCES:
- [Derived] Holmdahl V, Stark B, Clay L, Gunnarsson U, Strigard K. Long-term follow-up of full-thickness skin grafting in giant incisional hernia repair: a randomised controlled trial. Hernia. 2022 Apr;26(2):473-479. doi: 10.1007/s10029-021-02544-z. Epub 2021 Dec 14. PMID 34905143
- [Derived] Clay L, Stark B, Gunnarsson U, Strigard K. Full-thickness skin graft vs. synthetic mesh in the repair of giant incisional hernia: a randomized controlled multicenter study. Hernia. 2018 Apr;22(2):325-332. doi: 10.1007/s10029-017-1712-x. Epub 2017 Dec 15. PMID 29247365